CLINICAL TRIAL: NCT06338748
Title: Accuracy of the Dexcom G7 Continuous Glucose Monitoring System Following Cardiac Surgery
Acronym: DexcomG7
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24-157
Record Dates: First submitted 2024-03-23; First posted 2024-04-01 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Continuous Glucose Monitoring
MeSH Terms: interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Intervention Model Description: Patients undergoing heart surgery at the Cleveland Clinic (main campus) who would normally be tested for high sugar levels by poking a finger and using a test strip.
Masking Description: The study will involve using blinded Dexcom G7 continuous glucose monitoring (CGM) devices
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm (Other): All patients will receive the Dexcom G7 continuous glucose monitor (CGM)
  Interventions: Device: Continuous glucose monitor (CGM) Dexcom G7 used in blinded mode

INTERVENTIONS:
Device: Continuous glucose monitor (CGM) Dexcom G7 used in blinded mode — Dexcom G7 used in blinded mode

SUMMARY:
This is a prospective longitudinal study to study the agreement between a continuous glucose monitoring system (CGMS) versus current blood glucose monitoring. Subjects in this study will have their blood glucose measured regularly every 1-3 hours with current methods in the Cardiovascular Intensive Care Unit (CVICU), and by Point of Care (POC) fingerstick glucose using the Accucheck Inform II on the regular floors, and the CGMS reading at the same time will be captured. Subjects will have measurements taken throughout their stay in the CVICU and on the regular floors. Agreement and correlation between systems, as well as errors, will be calculated.

DETAILED DESCRIPTION:
The Dexcom G7 will be placed either by an anesthesiologist or nurse anesthetist, or critical care physician, nurse or nurse manager upon arrival to CVICU, post cardiac surgery.

Standard of care:

Accuchek will be done per standard of care for post operative patients that are in ICU

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old and above
* Planned cardiothoracic surgery
* Planned admission to Cleveland Clinic Main Campus building J5 or J6 or Q5 cardiovascular intensive care unit (CVICU) followed by transfer to the step down unit
* With or without known diabetes (as 75% of patients entering the CVICU have hyperglycemia requiring intravenous insulin infusion)
* If with known diagnosis of diabetes, diabetes can be type 1, type 2, or secondary (such as due to glucocorticoids or pancreatitis

Exclusion Criteria:

* Allergy to the material of the continuous glucose monitoring systems (CGMS) or the adhesive to be used
* Skin conditions precluding the use of the CGMS
* Pregnancy
* Other conditions that the investigators deem inappropriate for the study
* Patients receiving mechanical circulatory assist devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-11-02 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Compare accuracy of glucose readings obtained from Dexcom G7 compared to blood glucose obtained from arterial blood gas (ABG) or peripheral/central venous catheter or fingerstick point of care (POC) while patients are in the CVICU | 1 - 10 days
  Compare accuracy of glucose readings obtained from Dexcom G7 Compared to blood glucose obtained from arterial blood gas (ABG) or peripheral/central venous catheter or fingerstick POC while patients are in the CVICU
Compare accuracy of glucose readings obtained from Dexcom G7 compared to blood glucose obtained from fingerstick POC glucose when patients are on the regular floors | 1 - 10 days
  Compare accuracy of glucose readings obtained from Dexcom G7 compared to blood glucose obtained from fingerstick POC glucose when patients are on the regular floors

CONTACTS AND LOCATIONS:
Overall Officials: Lansang Cecilia, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No